CLINICAL TRIAL: NCT01501110
Title: Evaluation of the Effects of N-acetylcysteine on Thyroid Hormone Levels in the Low T3 Syndrome
Brief Title: Effects of N-acetylcysteine on Low T3 Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Programa de pós-graduação em endocrinologia (Unknown)
Responsible Party: Principal Investigator, Josi Vidart, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110061
Record Dates: First submitted 2011-11-25; First posted 2011-12-29 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myocardial Infarction; Euthyroid Sick Syndrome; Ischemic Heart Disease
Keywords: Euthyroid Sick Syndrome; low T3 syndrome; deiodases; oxidative stress; ischemic heart disease
MeSH Terms: conditions — Euthyroid Sick Syndromes; Myocardial Ischemia | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-acetylcysteine (Active Comparator): intra-venous infusion of 1200 mg of n-acetylcysteine twice a day for 48 hours.
  Interventions: Drug: N-acetylcysteine
- no intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: N-acetylcysteine — in infusion of 1200 mg of n-acetylcysteine twice a day for 48 hours
  Other Names: NAC; acetylcysteine
  Arms: n-acetylcysteine

SUMMARY:
The propose of this study is to determine whether N-acetylcysteine is effective in reversing the changes in thyroid hormones seen in critical illness, known as the low T3 syndrome.

DETAILED DESCRIPTION:
The low T3 syndrome or nonthyroidal illness is characterized by low levels of T3, normal or high normal levels of rT3, low or normal levels of T4 and inappropriately normal or low levels of TSH. These changes affect up to 75% of patients and have prognostic implications.

Interleukin-6 (IL6) seems to have a causative role in the pathogenesis of nonthyroidal illness. There is evidence that the reduction in serum T3 was inversely associated with serum IL-6, while the rT3 have a positive association. The mechanism of action of cytokines on the metabolism of thyroid hormones has not been determined and the potential role of cytokines on the deiodases has been the focus of research.

In a cell culture model study, IL-6 was able to suppress the conversion of T4 to T3 by deiodases type 1 and 2 and stimulate the inactivation of T3 by deiodase type 3, a situation similar to nonthyroidal illness. The use of N-acetylcysteine prevented this alterations, been consistent with the hypothesis that IL6 inhibits the function of the deiodases by increasing the oxygen reactive species and by consuming gluthathione or some gluthathione dependent cofactor.

Considering the absence of human studies evaluating the use of N-acetylcysteine in nonthyroidal illness, the aim of this study is to investigate whether NAC has in vivo effect on changes of thyroid hormones.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute myocardial infarction with less than 12 hours of evolution
* reperfusion therapy (primary angioplasty)

Exclusion Criteria:

* Thyroid disease
* Chronic renal disease with renal replacement therapy
* hepatic insufficiency
* immunosuppression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josi Vidart, Principal Investigator — Federal University of Rio Grande do Sul; Ana maia, Study Director — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Wajner SM, Goemann IM, Bueno AL, Larsen PR, Maia AL. IL-6 promotes nonthyroidal illness syndrome by blocking thyroxine activation while promoting thyroid hormone inactivation in human cells. J Clin Invest. 2011 May;121(5):1834-45. doi: 10.1172/JCI44678. Epub 2011 Apr 11. PMID 21540553
- [Background] Boelen A, Kwakkel J, Fliers E. Beyond low plasma T3: local thyroid hormone metabolism during inflammation and infection. Endocr Rev. 2011 Oct;32(5):670-93. doi: 10.1210/er.2011-0007. Epub 2011 Jul 26. PMID 21791567
- [Background] Maia AL, Goemann IM, Meyer EL, Wajner SM. Deiodinases: the balance of thyroid hormone: type 1 iodothyronine deiodinase in human physiology and disease. J Endocrinol. 2011 Jun;209(3):283-97. doi: 10.1530/JOE-10-0481. Epub 2011 Mar 17. PMID 21415143
- [Background] Bello G, Pennisi MA, Montini L, Silva S, Maviglia R, Cavallaro F, Bianchi A, De Marinis L, Antonelli M. Nonthyroidal illness syndrome and prolonged mechanical ventilation in patients admitted to the ICU. Chest. 2009 Jun;135(6):1448-1454. doi: 10.1378/chest.08-1816. Epub 2009 Mar 2. PMID 19255297
- [Background] Koenig RJ. Modeling the nonthyroidal illness syndrome. Curr Opin Endocrinol Diabetes Obes. 2008 Oct;15(5):466-9. doi: 10.1097/MED.0b013e32830eb838. PMID 18769221
- [Derived] Vidart J, Wajner SM, Leite RS, Manica A, Schaan BD, Larsen PR, Maia AL. N-acetylcysteine administration prevents nonthyroidal illness syndrome in patients with acute myocardial infarction: a randomized clinical trial. J Clin Endocrinol Metab. 2014 Dec;99(12):4537-45. doi: 10.1210/jc.2014-2192. PMID 25148231
- See also: Information on euthyroid sick syndrome — http://emedicine.medscape.com/article/118651-overview

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients with a diagnosis of acute myocardial infarction within 12 hours of evolution who underwent primary percutaneous coronary intervention and were admitted to the emergency and intensive care units of two tertiary hospitals in southern Brazil were recruited.
Pre-assignment Details: From the 83 patients enrolled, 15 met one of the following pre-established exclusion criteria: age younger than 18 or older than 80 yrs; primary thyroid disease; use of corticosteroids; chronic renal failure; severe hepatic insufficiency; severe immunosuppression; pregnant women or women undergoing postmenopausal hormone replacement.
Groups:
- no Intervention: No intervention / usual care
Period: Overall Study
Arm/Group | N-acetylcysteine | no Intervention
Started | 34 | 34
Completed | 34 | 33
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | no Intervention | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.4) | 57.4 (8.4) | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 27 | 24 | 51
Region of Enrollment [Number; unit: participants]
  Brazil | 34 | 33 | 67
TSH [Mean (Standard Deviation); unit: mcIU/mL] | 1.7 (1.2) | 1.6 (1.1) | 1.6 (1.2)
T3 [Mean (Standard Deviation); unit: ng/dL] | 100.4 (16.5) | 98.7 (20.7) | 99.3 (17.4)
T4 [Median (Standard Deviation); unit: mcg/dL] | 7.4 (1.9) | 7.4 (1.4) | 7.4 (1.5)
FT4 [Mean (Standard Deviation); unit: ng/dL] | 1.1 (0.2) | 1.1 (0.3) | 1.1 (0.2)
rT3 [Mean (Standard Deviation); unit: ng/dL] | 54.7 (8.1) | 55.2 (6.1) | 55 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Serum T3 Levels at 48 Hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | N-acetylcysteine | no Intervention
Number analyzed (Participants) | 34 | 33
ng/dL | 93.5 (20.1) | 96.5 (20.2)

ADVERSE EVENTS:
Time Frame: Adverse reactions were collected during drug infusion period (48 hours)
Arm/Group | N-acetylcysteine | no Intervention
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No